CLINICAL TRIAL: NCT06293456
Title: An Open Trial of a Novel Poetic Dignity Therapy Intervention to Enhance Meaning and Purpose for Sexual and Gender Minority Patients With Cancer
Brief Title: Study of Poetic Dignity Therapy for Sexual and Gender Minority Patients With Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-360
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: End of Life
Keywords: Dignity Therapy (DT); End of Life (EOL)
MeSH Terms: conditions — Death | interventions — Dignity Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dignity Therapy (Experimental): The DT intervention is a 45-75-minute virtual interview, which is recorded and transcribed within 1-2 weeks of the interview.
  Interventions: Other: Dignity Therapy

INTERVENTIONS:
Other: Dignity Therapy — A trained research staff member will conduct the DT interview virtually. The interview will occur or by phone only if the participant lacks access to technology for videoconferencing. The interviewer asks a series of open-ended questions that encourages patients to talk about their lives and what matters most to them.

SUMMARY:
The purpose of this study is to find out if dignity therapy is practical and works well for sexual and gender minority (SGM) patients in MSK. SGM includes, but is not limited to, people who identify as lesbian, gay, bisexual, transgender, and/or queer/questioning (LGBTQ+). Dignity therapy is a type of psychotherapy where the clinician asks the patient questions to allow the patient to express their individual life story and ultimately be able to create a legacy document of their experiences that can be shared with their loved ones.

ELIGIBILITY:
Inclusion Criteria:

* SGM (as per self-report) palliative care patients identified through Memorial Sloan Kettering Cancer Center's Palliative Care team and primary solid tumor oncology clinics.
* Age 18 and older (as per self-report/EHR)
* English-speaking as per the English language assessment items below and wil ing to receive the intervention in English.

  o What is the participant's preferred language?
* (Specify Lang)___________________________

  * How well does the participant speak English?
  * Very well (PARTICIPANT IS ELIGIBLE)
  * Well (PARTICIPANT is ELIGIBLE)
  * Not well (PARTICIPANT is NOT ELIGIBLE)
  * Not at all (PARTICIPANT is NOT ELIGIBLE)

Exclusion Criteria:

* Delirium/ altered mental status prohibitive of providing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
the number of patients who complete the intervention | 1 year
  This requires meeting both of the following criteria: i) collection of the DT Interview for 30 patients; and ii) delivery of the poem to at least 22 (>75%) participants.

CONTACTS AND LOCATIONS:
Overall Officials: William E Rosa, Ph.D., MBE, NP, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm